CLINICAL TRIAL: NCT01735071
Title: Multicenter, Randomized, Non-comparative, Phase II Trial on the Efficacy and Safety of the Combination of Bevacizumab and Trabectedin With or Without Carboplatin in Adult Women With Platinum Partially Sensitive Recurring Ovarian Cancer.
Brief Title: Bevacizumab and Trabectedin +/- Carboplatin in Advanced Ovarian Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mario Negri Institute for Pharmacological Research (Other)
Collaborators: PharmaMar (Industry); Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRFMN-OVA-6152
Record Dates: First submitted 2012-11-13; First posted 2012-11-28 (Estimated); Last update posted 2019-11-19 (Actual); Status verified 2019-11

CONDITIONS: Ovarian Epithelial Cancer Recurrent
Keywords: ovarian cancer; bevacizumab; trabectedin; carboplatin; randomized trial; phase II
MeSH Terms: conditions — Ovarian Neoplasms | interventions — Bevacizumab; Trabectedin; Carboplatin

STUDY DESIGN:
Intervention Model Description: This is a multicentre, randomized, non-comparative phase II study aimed at assessing efficacy and safety of two regimens according to a Bryant and Day two-stage design
Oversight: Data Monitoring Committee: No

ARMS (2):
- bevacizumab and trabectedin (Experimental): Arm A: bevacizumab (15 mg/kg) given as 1 hour infusion will be followed by trabectedin (1.1 mg/sqm) 3 hour iv infusion; to be repeated every 21 days until progression, unacceptable toxicity, patient or physician decision to discontinue, or death patients
  Interventions: Drug: bevacizumab and trabectedin
- bevacizumab, trabectedin and carboplatin (Experimental): Arm B: cycle 1-6, bevacizumab given as 1 hour infusion will be followed by carboplatin area under curve 4 (AUC 4) and trabectedin 3 hour iv infusion.
  Cycle 7- end of treatment, bevacizumab given as 1 hour infusion will be followed by trabectedin 3 hour iv infusion.
  Patient enrolled in arm B will receive (cycle 1-6): trabectedin 0.8 mg/m2 ,carboplatin AUC 4 day 1 every 28 days and bevacizumab 10 mg/kg iv on day 1 and day 15.
  From cycle 7 to disease progression, unacceptable toxicity, patient or physician decision to discontinue, or death patients will receive bevacizumab 15 mg/kg iv and trabectedin 1.1 mg/m2 day 1 every 21 days
  Interventions: Drug: bevacizumab, trabectedin and carboplatin

INTERVENTIONS:
Drug: bevacizumab and trabectedin — Arm A: bevacizumab (15 mg/kg) given as 1 hour infusion will be followed by trabectedin (1.1 mg/sqm) 3 hour iv infusion; to be repeated every 21 days until progression, unacceptable toxicity, patient or physician decision to discontinue, or death patients
  Other Names: Avastin; Yondelis
  Arms: bevacizumab and trabectedin
Drug: bevacizumab, trabectedin and carboplatin — Arm B: cycle 1- 6, bevacizumab given as 1 hour infusion will be followed by carboplatin AUC 4 and trabectedin 3 hour iv infusion.
  Cycle 7- end of treatment, bevacizumab given as 1 hour infusion will be followed by trabectedin 3 hour iv infusion.
  Patient enrolled in arm B will receive (cycle 1-6): trabectedin 0.8 mg/m2 ,carboplatin AUC 4 day 1 every 28 days and bevacizumab 10 mg/kg iv on day 1 and day 15.
  From cycle 7 to disease progression, unacceptable toxicity, patient or physician decision to discontinue, or death patients will receive bevacizumab 15 mg/kg iv and trabectedin 1.1 mg/m2 day 1 every 21 days
  Other Names: Avastin; Yondelis; Carboplatin
  Arms: bevacizumab, trabectedin and carboplatin

SUMMARY:
This study is aimed at assessing the efficacy and the safety of the combination of bevacizumab and trabectedin with or without carboplatin in adult women with epithelial ovarian cancer at first recurrence occurred 6-12 months after the end of the last (first or second) platinum-containing regimen. According to the Bryant and Day design the primary endpoints will be the proportion of progression-free patients at 6 months for the efficacy, and the proportion of patients with severe toxicity for the safety at the same time-point.

ELIGIBILITY:
Inclusion Criteria:

* Age≥18years
* Eastern Cooperative Oncology Group (ECOG)- performance status 0-2
* Cytological/histological diagnosis of epithelial ovarian cancer
* Progression free interval between 6-12 months (calculated from the first day of the last cycle of the previous last platinum-based chemotherapy until the date of progression confirmation through radiologic imaging)
* One or two previous platinum-based chemotherapy lines
* Measurable disease according to RECIST version 1.1
* Life expectancy ≥ 12 weeks
* Patients must be able to receive dexamethasone or its equivalent, as a premedication for trabectedin
* Written informed consents given before the enrolment according to International Conference on Harmonization/ Good Clinical Practice (ICH/GCP).

Exclusion Criteria:

* Prior treatment with trabectedin
* Prior progression while on therapy containing bevacizumab or other vascular endothelial growth factor (VEGF) pathway-target therapy
* Pre-existing grade > 1 sensitive/motor neurologic disorder
* Current or recent (within 30 days of first study dosing) treatment with another investigational drug
* Surgery (including open biopsy) within 4 weeks prior to the first planned dose of bevacizumab
* Current or recent (within 10 days prior to the first study drug dose) use of full-dose oral or parenteral anticoagulant or thrombolytic agent for therapeutic purposes (except for line patency, in which case international normalized ratio (INR) must be maintained below 1.5). Post operative prophylaxis with low molecular weight heparin sc is allowed
* Inadequate bone marrow function: absolute neutrophil count (ANC): <1.5 x 109/l, or platelet count <100 x 109/l or haemoglobin <9 g/dl. Patients may be transfused to maintain haemoglobin values ≥9 g/dl
* Inadequate coagulation parameters: activated partial thromboplastin time (APTT) >1.5 x upper limit of normal (ULN) or INR >1.5
* Inadequate liver function, defined as: serum (total) bilirubin > ULN for the institution AST/serum glutamic-oxaloacetic transaminase (SGOT) or ALT/ serum glutamic-pyruvic transaminase (SGPT) >2.5 x ULN
* Inadequate renal function: serum creatinine >1.5 mg/dL or >132 micromol/L and urine dipstick for proteinuria > or = 2+ and >1g of protein in their 24-hour urine collection
* History or evidence of brain metastases or spinal cord compression
* Pregnant, breastfeeding women and women of child bearing potential, who do not agree to use a medically acceptable method of contraception through the treatment period and for 6 months after discontinuation of treatment
* History or evidence of thrombotic or hemorrhagic disorders; including cerebrovascular accident, stroke or transient ischemic attack or sub-arachnoid haemorrhage within 6 months prior to the first study treatment
* Uncontrolled hypertension (sustained systolic >150 mmHg and/or diastolic >100 mmHg despite antihypertensive therapy) or clinically significant (i.e. active) cardiovascular disease, including: myocardial infarction or unstable angina within 6 months prior to the first study treatment, New York Heart Association grade II or greater congestive heart failure, serious cardiac arrhythmia requiring medication
* History of bowel obstruction, including subocclusive disease, related to the underlying disease and history of abdominal fistula, gastrointestinal perforation or intra-abdominal abscess. Evidence of recto-sigmoid involvement by pelvic examination or bowel involvement on CT scan or clinical symptoms of bowel obstruction
* Non-healing wound, ulcer or bone fracture
* hepatitis C virus (HCV) positivity
* Other malignancy within the last 5 years, except for adequately treated carcinoma in situ of the cervix or squamous carcinoma of the skin, or adequately controlled limited basal cell skin cancer.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2013-07 (Actual); Primary Completion 2018-03-18 (Actual); Study Completion 2018-03-18 (Actual)

PRIMARY OUTCOMES:
Progression Free Survival at 6 months (PFS-6) | from randomization up to 6 months
  The PFS-6, defined as the percentage of patients who are alive and progression free at 6 months after the randomization.
Proportion of patients with severe toxicity within 6 months from randomization. | from randomization up to 6 months
  The following conditions will be considered as severe toxicity:
  * absolute neutrophil count (ANC) < 0.5x109/L lasting > 7 days and/or with fever
  * platelets < 25x109/L
  * any other grade 3-4 (evaluated by the National Cancer Institute-Common Terminology Criteria for Adverse Events [NCI-CTCAE] version 4.0) non-hematological toxicities except for reversible nausea/vomiting, diarrhea, hypersensitivity reactions, and alanine aminotransferase (ALT) or aspartate aminotransferase (AST) elevation reversible to grade 1 by day 28
  * any toxicity causing a delay of >14 days in the following cycle

SECONDARY OUTCOMES:
Progression Free Survival (PFS) | from randomization up to 30 months
  Defined for each patient as the time from the date of randomization to the date of first progression, second primary malignancy or death for any cause, whichever comes first. Subjects not progressed or died at the time of the analysis will be censored at the last disease assessment date.
Overall survival at 12 months (OS-12) | one year
  Defined as the percentage of patients who are alive at 12 months after the randomization.
Clinical Benefit (CB) | from randomization up to 30 months
  clinical benefit, defined as the percentage of patients who are judged by the Investigators to have a complete response (CR), or partial response (PR) or stable disease (SD) according to the Response Evaluation Criteria In Solid Tumors (RECIST) criteria, version 1.1 after 12 weeks from the date of randomization.
Incidence of Adverse Events (AEs) | from randomization up to 30 months
  Incidence of AEs, according to NCI-CTCAE, version 4.0
Maximum toxicity grade | from randomization up to 30 months
  Maximum toxicity grade experienced by each patient for each specific toxicity
Percentage of patients experiencing grade 3-4 toxicity for each specific toxicity | from randomization up to 30 months
  Percentage of patients experiencing grade 3-4 toxicity for each specific toxicity during the study
Patients with at least a Serious Adverse Drug Reaction (SADR) | from randomization up to 30 months
  Patients with at least a SADR during the study
Patients with at least a Suspect Unexpected Serious Adverse Reaction (SUSAR). | from randomization up to 30 months
  Patients with at least a suspect unexpected serious adverse reaction during the study
Percentage of patients with dose and/or time modifications | from randomization up to 30 months
  Percentage of patients with dose and/or time modifications of the study drugs
Percentage of premature withdrawals | from randomization up to 30 months
  Percentage of premature withdrawals of the enrolled patients
Patients with at least a Serious Adverse Event (SAE) | from randomization up to 30 months
  Patients with at least a SAE during the study
Nature of AEs | from randomization up to 30 months
  Nature of AEs, according to NCI-CTCAE, version 4.0
Severity of AEs | from randomization up to 30 months
  Severity of AEs, according to NCI-CTCAE, version 4.0
Seriousness of AEs | from randomization up to 30 months
  Seriousness of AEs according to NCI-CTCAE, version 4.0

CONTACTS AND LOCATIONS:
Overall Officials: Nicoletta Colombo, Medical D, Principal Investigator — IRCCS Istituto Europeo di Oncologia di Milano
Locations (7):
- Italy (7):
  - Azienda Ospedaliera Spedali Civili di Brescia, Brescia
  - Istituto Europeo di Oncologia, Milan
  - AO Fatebenefratelli e Oftalmico, Milan
  - Azienda Ospedaliera S. Gerardo, Monza
  - Istituto Oncologico Veneto, Padua
  - Policlinico Universitario Agostino Gemelli di Roma, Roma
  - Mauriziano Hospital, Torino

REFERENCES:
- [Result] Colombo N, Zaccarelli E, Baldoni A, Frezzini S, Scambia G, Palluzzi E, Tognon G, Lissoni AA, Rubino D, Ferrero A, Farina G, Negri E, Pesenti Gritti A, Galli F, Biagioli E, Rulli E, Poli D, Gerardi C, Torri V, Fossati R, D'Incalci M. Multicenter, randomised, open-label, non-comparative phase 2 trial on the efficacy and safety of the combination of bevacizumab and trabectedin with or without carboplatin in women with partially platinum-sensitive recurrent ovarian cancer. Br J Cancer. 2019 Oct;121(9):744-750. doi: 10.1038/s41416-019-0584-5. Epub 2019 Sep 20. PMID 31537908